CLINICAL TRIAL: NCT03351218
Title: Neuronal Correlates of Agency in Dystonia
Brief Title: Agency in Dystonia
Acronym: AGENT10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C17-04; 2017-A01231-52 (Registry Identifier: RCB)
Record Dates: First submitted 2017-10-10; First posted 2017-11-22 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-03

CONDITIONS: Dystonia, Primary
MeSH Terms: conditions — Dystonic Disorders

STUDY DESIGN:
Intervention Model Description: Two groups study : patients versus healthy controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Other): 25 patients with cervical and 25 patients with myoclonus dystonia
  Interventions: Behavioral: Behavioral testing - computerized tasks
- Controls (Other): 50 healthy volunteers matched to patents ( age, sex)
  Interventions: Behavioral: Behavioral testing - computerized tasks

INTERVENTIONS:
Behavioral: Behavioral testing - computerized tasks — Cognitive behavioral testing and cerebral MRI

SUMMARY:
In this study, using computerized cognitive assessments combined with multi-modal neuroimaging approach investigators aim to address three specific questions on patients with cervical and myoclonus dystonia:

(i) investigate various aspects of the sense of agency and relationship to the severity of dystonia symptoms, (ii) characterize the possible link between abnormalities of movement perception and alteration of sense of agency in dystonia, (iii) (identify the neuronal underpinnings of the defective sense of agency in dystonia.

DETAILED DESCRIPTION:
This is a single-centre, two-group ( dystonia and control), case-control study using behavioural and novel multimodal neuroimaging techniques to address the study aims.

The battery of the tasks will include explicit-agency tasks, a visual discrimination task on objects movement perception. The magnetic resonance acquisition protocol will include MP2RAGE structural (10 min duration), multi echo (3 echo times) multiband (MB factor 4) resting state functional neuroimaging (15 minutes duration) and multi shell diffusion imaging sequence (15 minutes duration)

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of isolated adult-onset cervical dystonia (CD) or myoclonus dystonia (MD);
* duration of disease of more than one year
* no botulinum toxin injection for at least three months before the study
* normal or corrected-to-normal vision.

Exclusion Criteria

* any neurological history except for dystonia,
* history of dopamine antagonist treatment,
* secondary dystonia,
* dystonia in the upper limbs,
* inability to maintain gaze straight.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
agency tasks behavioral outcome measures | throughout study completion, an average 2 years
  response time
agency tasks behavioral outcome measures | throughout study completion, an average 2 years
  response accuracy in tasks trials

SECONDARY OUTCOMES:
MRI measures | throughout study completion, an average 2 years
  cortical thickness
MRI measures | throughout study completion, an average 2 years
  basal ganglia volume

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'investigation Clinique, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Tarrano C, Lamy JC, Delorme C, McGovern EM, Atkinson-Clement C, Brochard V, Thobois S, Tranchant C, Grabli D, Degos B, Corvol JC, Pedespan JM, Krystkoviak P, Houeto JL, Degardin A, Defebvre L, Apartis E, Vidailhet M, Roze E, Worbe Y. Tactile Temporal Discrimination Is Impaired in Myoclonus-Dystonia. Mov Disord. 2020 Dec;35(12):2356-2357. doi: 10.1002/mds.28253. Epub 2020 Sep 22. No abstract available. PMID 32960985
- [Result] Tarrano C, Wattiez N, Delorme C, McGovern EM, Brochard V, Thobois S, Tranchant C, Grabli D, Degos B, Corvol JC, Pedespan JM, Krystkoviak P, Houeto JL, Degardin A, Defebvre L, Valabregue R, Vidailhet M, Pouget P, Roze E, Worbe Y. Visual sensory processing is altered in myoclonus dystonia. Mov Disord. 2020 Jan;35(1):151-160. doi: 10.1002/mds.27857. Epub 2019 Sep 30. PMID 31571302
- [Result] Zito GA, Tarrano C, Jegatheesan P, Ekmen A, Beranger B, Rebsamen M, Hubsch C, Sangla S, Bonnet C, Delorme C, Meneret A, Degos B, Bouquet F, Brissard MA, Vidailhet M, Gallea C, Roze E, Worbe Y. Somatotopy of cervical dystonia in motor-cerebellar networks: Evidence from resting state fMRI. Parkinsonism Relat Disord. 2022 Jan;94:30-36. doi: 10.1016/j.parkreldis.2021.11.034. Epub 2021 Nov 30. PMID 34875561
- [Result] Zito GA, Tarrano C, Ouarab S, Jegatheesan P, Ekmen A, Beranger B, Valabregue R, Hubsch C, Sangla S, Bonnet C, Delorme C, Meneret A, Degos B, Bouquet F, Apoil Brissard M, Vidailhet M, Hasboun D, Worbe Y, Roze E, Gallea C. Fixel-Based Analysis Reveals Whole-Brain White Matter Abnormalities in Cervical Dystonia. Mov Disord. 2023 Jul;38(7):1187-1196. doi: 10.1002/mds.29425. Epub 2023 May 6. PMID 37148555
- [Result] Zito GA, Roze E, Tarrano C, Ouarab S, Jegatheesan P, Ekmen A, Beranger B, Valabregue R, Hubsch C, Sangla S, Bonnet C, Delorme C, Meneret A, Degos B, Bouquet F, Apoil Brissard M, Vidailhet M, Hasboun D, Pouget P, Worbe Y, Gallea C. Abnormal Connectivity of the Head Neural Integrator in Cervical Dystonia. Mov Disord. 2025 Nov;40(11):2321-2330. doi: 10.1002/mds.70014. Epub 2025 Sep 5. PMID 40910449
- [Result] Atkinson-Clement C, Tarrano C, Porte CA, Wattiez N, Delorme C, McGovern EM, Brochard V, Thobois S, Tranchant C, Grabli D, Degos B, Corvol JC, Pedespan JM, Krystkoviak P, Houeto JL, Degardin A, Defebvre L, Valabregue R, Rosso C, Apartis E, Vidailhet M, Pouget P, Roze E, Worbe Y. Dissociation in reactive and proactive inhibitory control in Myoclonus dystonia. Sci Rep. 2020 Aug 18;10(1):13933. doi: 10.1038/s41598-020-70926-x. PMID 32811896